CLINICAL TRIAL: NCT01438580
Title: The Effect and Safety of Different Intensity Anticoagulation Therapy in Elderly Patients With Non-valvular Atrial Fibrillation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Wu Jun, First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30900602
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial ﬁbrillation; stroke; warfarin; aspirin
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Warfarin; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard intensity warfarin group (Experimental): Eligible 80 patients(83.14±4.05,33.0%)with chronic NVAF were randomly assigned to this group and the target international normalised ratio(INR) was 2.1-3.0
  Interventions: Drug: Warfarin
- low intensity warfarin group (Experimental): Eligible 81 patients(84.0±4.71,33.5%)with chronic NVAF were randomly assigned to this group and the target international normalised ratio(INR) was 1.5-2.0
  Interventions: Drug: Warfarin
- aspirin group (Active Comparator): Eligible 81 patients(83.4±5.13,33.5%)with chronic NVAF were randomly assigned to this group and 100mg aspirin was administrated every day
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: Warfarin — Patients randomised to receive warfarin were initiated on treatment at the baseline dose of 1.25mg daily and then gradually increase the amount to the target INR range.
  Arms: low intensity warfarin group; standard intensity warfarin group
Drug: aspirin — 100mg aspirin was administrated every day
  Arms: aspirin group

SUMMARY:
Current guidelines recommend standard warfarin anticoagulation international normalized ratio (INR) goal of 2.0-3.0 in adults with non valvular atrial fibrillation (NVAF). The investigators hypothesized that low-intensity warfarin (INR 1.5-2.0) has the same effectiveness and better security in elderly patients (>75) with NVAF.

DETAILED DESCRIPTION:
Atrial fibrillation is the commonest chronic arrhythmia in clinical practice, especially in octogenarians. Nonvalvular atrial ﬁbrillation increases the risk of ischemic stroke by approximately 5-fold and these strokes result in higher mortality and disability. Warfarin is recommended as ﬁrst line anticoagulation treatment in patients with NVAF who are at moderate or high risk of stroke,while antiplatelet agents, such as aspirin, give a more convenient but less effective alternative in the prevention of ischemic stroke and are recommended in low risk patients.Current guideline about warfarin anticoagulation therapy recommend that target INR value must be maintained between 2.0 and 3.0,which not only reduces the frequency of ischaemic stroke but also its low incidence of major bleeding. However, the current status of anticoagulation therapy for elderly Chinese AF patients, particularly in aged over 80 years, is not clear. The purpose of the present study was to test the hypothesis that an INR target of 1.5-2.0 can provide the same efficacy and better safety as compare with a standard target of 2.0-3.0 in patients over 75 with NVAF.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of atrial fibrillation
2. Echocardiography confirmed a non-valvular heart disease
3. Age≥75 years

Exclusion Criteria:

1. Unable to cooperate with doctors
2. Life expectancy of less than 1 year
3. Rheumatic heart disease or dilated cardiomyopathy
4. History of artificial valve replacement surgery
5. Infectious endocarditis
6. Stroke or transient ischemic attack(TIA) within the last 6 months
7. Previous history of intracranial hemorrhage, gastrointestinal, respiratory or urogenital bleeding
8. Previous intolerance/allergy to warfarin or aspirin
9. Blood pressure greater than 180/110 mmHg
10. Chronic liver dysfunction, alanine aminotransferase above the normal reference value of the upper limit 3 times
11. Chronic renal failure, serum creatinine clearance rate (Ccr) less than 30 ml / min
12. Patient was receiving antiplatelet or anticoagulant therapy due to other reasons

Ages: 75 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
major haemorrhage | 2 years
  Major haemorrhage was defined as intracranial hemorrhage, gastrointestinal bleeding, bleeding requiring hospitalization and surgical intervention, a reduction of hemoglobin by≥2 g/dL, requiring red blood cells transfusion ≥2 units.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. In addition, the number of bleeding events was recorded.
ischaemic stroke | 2 years
  ischaemic stroke was defined as a blockage in an artery that supplies blood to the brain , resulting in a deficiency in blood flow and focal neurological deficit lasting >24 hours.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. In addition, the number of ischaemic stroke was recorded.

SECONDARY OUTCOMES:
minor bleeding | 2.5years
  Minor bleeding was any other bleeding requiring modiﬁcation of the antithrombotic regimen,such as hematuria, gingival, conjunctival bleeding and so on.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. In addition, the number of minor bleedinge was recorded.
myocardial infarction | 2.5 years
  Myocardial infarction was defined as occurrence of typical chest pain, ECG and cardiac enzyme abnormalities.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. The number of myocardial infarction was recorded.
deep vein thrombosis | 2.5 years
  Deep vein thrombosis (DVT) was defined as a blood clot in a major vein that usually develops in the legs and/or pelvis and blocks blood flow, which can be diagnosised by ultrasound.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. The number of deep vein thrombosis was recorded.
pulmonary embolism | 2.5 years
  Pulmonary embolism was defined as occurrence of typical shortness of breath, chest pain, D-dimer and CT pulmonary angiography abnormalities.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. The number of pulmonary embolism was recorded.
cardiovascular death | 2.5 years
  Cardiovascular causes of death included myocardial infarction, heart failure, cardiac arrhythmia.
  Follow-up study visits were scheduled for once a week in the first month and then every 3 months. The number and results of INR tests, liver and kidney function tests were recorded. The number of cardiovascular death was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Guo Yan, doctor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Division of Geriatrics, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wu J, Wang J, Jiang S, Xu J, Di Q, Zhou C, Min X, Pang S, Wang H, Xu D, Guo Y. The efficacy and safety of low intensity warfarin therapy in Chinese elderly atrial fibrillation patients with high CHADS2 risk score. Int J Cardiol. 2013 Sep 10;167(6):3067-8. doi: 10.1016/j.ijcard.2012.11.078. Epub 2012 Nov 28. No abstract available. PMID 23200268